CLINICAL TRIAL: NCT00316147
Title: Phase IIIb, Open, Randomized, Multicenter Study to Assess the Immunogenicity & Safety of GSK Biologicals' Combined DTPa-HBV-IPV/Hib Vaccine in Indian Infants When Given at 6-10-14 Weeks of Age or at 2-4-6 Months of Age
Brief Title: Immunogenicity & Safety of GSK's Combined DTPa-HBV-IPV/Hib Vaccine in Indian Infants at 2 Diff Vaccination Schedules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104005
Record Dates: First submitted 2006-02-21; First posted 2006-04-20 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus; Haemophilus Influenzae Type b; Hepatitis B; Poliomyelitis
Keywords: diphtheria; tetanus; poliomyelitis; pertussis; hepatitis B; Prophylaxis; Haemophilus influenza type b diseases
MeSH Terms: conditions — Diphtheria; Tetanus; Haemophilus Infections; Hepatitis B; Poliomyelitis; Whooping Cough

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib vaccine

SUMMARY:
In this study, infants who were previously vaccinated with hepatitis B vaccine at birth will be randomly allocated into two groups:

* one group of subjects will receive diphtheria, tetanus, acellular pertussis- hepatitis B virus-inactivated poliovirus/Haemophilus influenzae type b (DTPa-HBV-IPV/Hib) vaccine at 6-10-14 weeks of age
* the second group of subjects will receive DTPa-HBV-IPV/Hib vaccine at 2-4-6 months of age

DETAILED DESCRIPTION:
DTPa-HBV-IPV/Hib vaccine will be administered at two schedules (i.e. 6-10-14 weeks of age OR 2-4-6 months of age) in infants who were previously vaccinated with hepatitis B vaccine at birth. The duration of the study will be approximately 3 months for each subject who will receive vaccination at 6-10-14 weeks of age and approximately 5 months for each subject who will receive vaccination at 2-4-6 months of age. Intervention name: Diphteria, tetanus, acellular pertussis, hepatitis B, poliovirus types 1, 2, 3 & Haemophilus influenzae type b vaccine

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female infant between, and including, 6 to 10 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Born after a normal gestation period (between 36 and 42 weeks).
* Should have received a birth dose of hepatitis B vaccine, as evidenced by vaccination/immunisation certificate.

Exclusion Criteria:

* Use of any investigational or non-registered product (vaccine or drug) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the first vaccine dose and ending 30 days after the last dose (with the exception of oral polio vaccine as a birth dose or for a pulse polio program, as per local, regional, or national requirements).
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis and Haemophilus influenzae type b diseases.
* Known exposure to diphtheria, tetanus, Bordetella pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b diseases since birth.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224
Dates: Start 2005-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
1M post-dose 3, vaccine response for pertussis and anti-poliovirus types 1, 2, and 3 titers

SECONDARY OUTCOMES:
1M post-dose 3, antibody levels against all antigens
After each dose, solicited (day 0-3, local and general) and unsolicited (day 0-30) events
Serious adverse events (SAEs) for entire study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Baroda
  - GSK Investigational Site, Goa
  - GSK Investigational Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register